CLINICAL TRIAL: NCT05677542
Title: Secukinumab (Cosentyx®) Effectiveness in Axial Spondyloarthritis and Psoriatic Arthritis Patients Using Artificial Intelligence (SpAINET): Spanish Multicenter, Retrospective, Real World Evidence Study
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457FES07
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Axial Spondyloarthritis; Psoriatic Arthritis
Keywords: Axial spondyloarthritis;; Psoriatic Arthritis;; electronic health records;; natural language processing;; artificial intelligence
MeSH Terms: conditions — Axial Spondyloarthritis; Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Axial Spondyloarthritis Patients: Patients with Axial Spondyloarthritis
  Interventions: Drug: secukinumab
- Psoriatic Arthritis Patients: Patients with Psoriatic Arthritis
  Interventions: Drug: secukinumab

INTERVENTIONS:
Drug: secukinumab — all patients who received secukinumab

SUMMARY:
This was a multicenter, retrospective, and non-interventional study using secondary data captured in the Electronic Health Records (EHRs). The extraction of the data captured in the EHRs was performed with EHRead® by SAVANA, an innovating data-driven system based on Natural Language Processing (NLP) and big data analytics. Data was extracted and analyzed at Index Date, Follow Up, or as specified for each variable.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* Diagnosed with axSpA or PsA.
* Had received or are receiving bDMARD, independently of the line of treatment, from January 2018 to data collection.
* Had at least 3 months follow up from first bDMARD administration.
* Patients with EHRs.

Exclusion Criteria:

• Receiving bDMARD within a clinical trial from January 2018 to data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a multicenter, retrospective, and non-interventional study using secondary data captured in the Electronic Health Records (EHRs).
Sampling Method: Non-Probability Sample
Enrollment: 758 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving disease control status at 6 months (±3 months) of secukinumab treatment | month 6
  Disease control was defined as:
  For Axial Spondyloarthritis (axSpA) population: Bath Ankylosing Spondylitis Functional Index (BASDAI) score < 4. If BASDAI was not available, Ankylosing Spondylitis Disease Activity Score (ASDAS) < 2.1 was used.
  For Psoriatic Arthritis (PsA) population: Disease Activity in PSoriatic Arthritis (DAPSA) score < 14. If DAPSA was not available, Disease activity score 28 (DAS-28) < 3.2 was used.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Spain (3):
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Valencia

IPD SHARING:
Plan to Share IPD: No